CLINICAL TRIAL: NCT04364438
Title: A Randomized Controlled Trial on Effectiveness of Electric Muscle Stimulation (EMS) and Transcutaneous Electric Nerve Stimulation (TENS) in Patients With Overactive Bladder
Brief Title: Effectiveness of EMS and TENS in Patients With Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Sajid rashid, Principal Investigator, Isra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1502-PhD-007
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Overactive Bladder
Keywords: Urinary Bladder, Overactive; Urinary Incontinence; Quality of Life; Transcutaneous Electric Nerve Stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The total sample will be divided into three groups i.e., Control group and two experimental groups. Control group will be treated with conventional medical treatment including anticholinergics and pelvic floor muscle exercises while 1st experimental group will be treated with conventional treatment and EMS and the 2nd experimental group will be treated with conventional treatment and TENS.
  initial results will be measured by Overactive Bladder Scoring System and King's Health Questionnaire. A follow up chart will be maintained after every 03 weeks regarding the symptoms of the patients and Quality of Life. After 12 weeks( completion of treatment) the patient will be re evaluated for their symptoms and graded by using Overactive Bladder Scoring System and King's Health Questionnaire.
  A comparison will be made among data obtained from 03 groups to check the effectiveness of intervention by using statistical analysis
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Patients will be treated with conventional medical treatment for overactive bladder including anticholinergic drugs and pelvic floor muscle exercises
- EMS Group (Experimental): Patients will be treated with conventional medical treatment for overactive bladder including anticholinergic drugs and pelvic floor muscle exercises along with Electric Muscle Stimulation (EMS)
  Interventions: Device: Electric Muscle Stimulation
- TENS Group (Experimental): Patients will be treated with conventional medical treatment for overactive bladder including anticholinergic drugs and pelvic floor muscle exercises along with Transcutaneous Electric Nerve Stimulation (TENS)
  Interventions: Device: Transcutaneous Electric Nerve Stimulation

INTERVENTIONS:
Device: Electric Muscle Stimulation — EMS is believed to produce some inhibition of the bladder, allowing the bladder to reach a greater volume. This is believed to occur because electrical stimulation also stimulates nerves in the pelvic floor. In most people, bladder voiding is inhibited when the skin of the pelvis is touched or otherwise manipulated. This inhibition is via a reflex in the spinal cord that may have evolved to inhibit voiding during sexual contact. The pelvic floor nerves are responsible for transmitting the sensation of touch from the pelvis to the spinal cord. Electrical stimulation of these nerves thus activates sensory fibers that cause inhibition of bladder voiding via a reflex mechanism in the spinal cord. This may explain EMS is an effective treatment for people with incontinence.
  Other Names: EMS
  Arms: EMS Group
Device: Transcutaneous Electric Nerve Stimulation — TENS is based on the gate control theory of abolishing the local micturition reflex arc. It is a non-pharmacological method of inhibiting the presynaptic afferent neurons carrying impulses from bladder by stimulating the nerves of peripheral segmental dermatome (gate control theory of electro modulation by stimulating the peripheral nerves corresponding to the visceral organ). It acts at the level of primitive voiding reflex coordinating the bladder, sphincter and the pelvic floor. Detrusor hyperreflexia can be inhibited by direct inhibition of impulses in the preganglionic afferent neuron or by inhibition of bladder preganglionic neurons of the efferent limb of micturition reflex.
  Other Names: TENS
  Arms: TENS Group

SUMMARY:
Overactive bladder (OAB) syndrome is a well-recognized set of symptoms which patient experience during the storage phase of the micturition cycle. It is characterized by urgency (a sudden compelling desire to pass urine which is difficult to defer) which, in almost all patients, is accompanied by increased frequency and nocturia and, particularly in female patients, by urgency incontinence.

DETAILED DESCRIPTION:
Leaking urine is called "incontinence". Stress urinary incontinence (SUI), is another common bladder problem. It's different from OAB. People with SUI leak urine while sneezing, laughing or doing other physical activities. If you have an overactive bladder, you may feel embarrassed, isolate yourself, or limit your work and social life.

Overactive bladder (OAB) is a very common clinical condition, with an overall prevalence estimated at 11.5% in the general population of Pakistan.

In traditional medicine and recent years, nerve stimulation has been introduced as a replacement therapy for managing several disorders such as overactive bladder. However, there is still controversy in this regard. Therefore, the present study is aimed to find out the effectiveness of Electric Muscle Stimulation and Transcutaneous Electric Nerve Stimulation in treatment of overactive bladder.To overcome this controversy we need to do this study in Pakistan and find out whether there is any role of EMS and TENS in the management of OAB.

OAB is one of the important conditions that lead to the limitation in activity and participation due to dribbling, urgency and frequency of urination. According to literature review there is a strong linkage between OAB rehabilitation and improvement of patient symptoms. The Neuromodulation plays a significant role in the management of OAB. The proper task specific rehabilitation not only improves the functional status of a person rather it enhances the quality of life and their active role in community. In routine rehabilitation main focus is always on the role of pelvic floor exercises but Neuromodulation is still neglected in treatment regimen of OAB in Pakistan. The patients will profit in better help of manifestations if Neuromodulation intervention is applied that is upheld by proof for the treatment of OAB. The consequences of the investigation will be useful for the Physical Therapists in planning and picking best treatment approach for the treatment of OAB.

TENS is based on the gate control theory of abolishing the local micturition reflex arc. It is a non-pharmacological method of inhibiting the presynaptic afferent neurons carrying impulses from bladder by stimulating the nerves of peripheral segmental dermatome (gate control theory of electro modulation by stimulating the peripheral nerves corresponding to the visceral organ). It acts at the level of primitive voiding reflex coordinating the bladder, sphincter and the pelvic floor. Detrusor hyperreflexia can be inhibited by direct inhibition of impulses in the preganglionic afferent neuron or by inhibition of bladder preganglionic neurons of the efferent limb of micturition reflex.

EMS is also believed to produce some inhibition of the bladder, allowing the bladder to reach a greater volume. This is believed to occur because electrical stimulation also stimulates nerves in the pelvic floor. In most people, bladder voiding is inhibited when the skin of the pelvis is touched or otherwise manipulated. This inhibition is via a reflex in the spinal cord that may have evolved to inhibit voiding during sexual contact. The pelvic floor nerves are responsible for transmitting the sensation of touch from the pelvis to the spinal cord. Electrical stimulation of these nerves thus activates sensory fibers that cause inhibition of bladder voiding via a reflex mechanism in the spinal cord. This may explain EMS is an effective treatment for people with incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female patients ≥35years to 60 years with OAB symptoms of urgency, frequency, nocturia and urgency urinary incontinence (UUI).8
* Those who have symptoms of urinary frequency and urgency lasting more than 3 months.
* Those who have an average urinary frequency of more than eight times per day and urgency defined by the urgency rating scale (URS) on the bladder diary of more than 2 points. 9

Exclusion Criteria:

* Diagnosed with Urinary Tract Infection by urine examination.
* Stress urinary incontinence without symptoms of OAB.
* History of cystocele, uterine prolapse or similar condition.
* History of obstructive uropathy such as urinary stones and urinary tumors.
* Prostate
* Malignancy

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Scoring System (Change is being assessed) | Baseline and week 12
  The Overactive Bladder Scoring System is a symptom assessment questionnaire designed to quantify OAB symptoms into a single score. The questionnaire consists of 4 questions on OAB symptoms with maximum scores ranging from 2 to 5: daytime frequency (2 points), night-time frequency (3 points), urgency (5 points), and UUI (5 points). The total score ranges from 0 to 15 points, with higher scores indicating higher symptom severity. Initial results will be measured by using overactive bladder scoring system. After 12 weeks ( Completion of Treatment) patients will be re evaluated for their symptoms and graded again by using overactive bladder scoring system. A comparison will be made among data obtained from 03 groups to check the effectiveness of intervention

SECONDARY OUTCOMES:
King's Health Questionnaire (Change is being assessed) | Baseline and week 12
  The King's Health Questionnaire (KHQ) is a disease-specific health-related quality-of-life (HRQoL) instrument to measure HRQoL of patients with urinary incontinence. Since its development the KHQ has been widely used in clinical studies as a valid, reliable and clinically sensitive endpoint. The individual items in the domains are scaled from 0 ( Best) to 100 ( Worst).

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Babur, Ph.D, Study Chair — Isra University, Islamabad
Locations (1):
- Sajid Rashid, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacDiarmid SA, Peters KM, Shobeiri SA, Wooldridge LS, Rovner ES, Leong FC, Siegel SW, Tate SB, Feagins BA. Long-term durability of percutaneous tibial nerve stimulation for the treatment of overactive bladder. J Urol. 2010 Jan;183(1):234-40. doi: 10.1016/j.juro.2009.08.160. PMID 19913821
- [Background] Preyer O, Umek W, Laml T, Bjelic-Radisic V, Gabriel B, Mittlboeck M, Hanzal E. Percutaneous tibial nerve stimulation versus tolterodine for overactive bladder in women: a randomised controlled trial. Eur J Obstet Gynecol Reprod Biol. 2015 Aug;191:51-6. doi: 10.1016/j.ejogrb.2015.05.014. Epub 2015 Jun 3. PMID 26073262
- [Background] Jokhio AH, Rizvi RM, Rizvi J, MacArthur C. Urinary incontinence in women in rural Pakistan: prevalence, severity, associated factors and impact on life. BJOG. 2013 Jan;120(2):180-186. doi: 10.1111/1471-0528.12074. PMID 23240797
- [Background] Sharma N, Rekha K, Srinivasan KJ. Efficacy of Transcutaneous Electrical Nerve Stimulation in the Treatment of Overactive Bladder. J Clin Diagn Res. 2016 Oct;10(10):QC17-QC20. doi: 10.7860/JCDR/2016/21683.8729. Epub 2016 Oct 1. PMID 27891403
- [Background] Janssen DA, Martens FM, de Wall LL, van Breda HM, Heesakkers JP. Clinical utility of neurostimulation devices in the treatment of overactive bladder: current perspectives. Med Devices (Auckl). 2017 Jun 1;10:109-122. doi: 10.2147/MDER.S115678. eCollection 2017. PMID 28615976
- [Background] Sensoy N, Dogan N, Ozek B, Karaaslan L. Urinary incontinence in women: prevalence rates, risk factors and impact on quality of life. Pak J Med Sci. 2013 May;29(3):818-22. doi: 10.12669/pjms.293.3404. PMID 24353635
- [Background] Badia Llach X, Castro Diaz D, Conejero Sugranes J. [Validity of the King's Health questionnaire in the assessment of quality of life of patients with urinary incontinence. The King's Group]. Med Clin (Barc). 2000 May 6;114(17):647-52. doi: 10.1016/s0025-7753(00)71390-x. Spanish. PMID 10900603
- See also: The Effect of Electrical Nerve Stimulation in Management of — https://www.sid.ir/FileServer/JE/5074020171248.pdf
- See also: Method to control an overactive bladder — https://patentimages.storage.googleapis.com/46/03/59/1de87a2e1f5ba6/US6836684.pdf
- See also: Describing bladder storage function: overactive bladder syndrome and detrusor overactivity — https://doi.org/10.1016/j.urology.2003.09.050